CLINICAL TRIAL: NCT01386138
Title: Treating South African Pregnant Women for Methamphetamine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DA030565
Record Dates: First submitted 2011-06-29; First posted 2011-06-30 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: HIV; Drug Addiction
Keywords: HIV; HIV Risk; Sexually Transmitted Infections; Women; Pregnancy; Neonatal Health; Drug Use; Drug Treatment; Gender-specific Treatment; Methamphetamine; Opioids; Cocaine; Injection Drugs; Stimulants; Alcohol; Mandrax; Marijuana; Nicotine
MeSH Terms: conditions — Substance-Related Disorders; Sexually Transmitted Diseases; Marijuana Abuse

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RBT+WHIC (Experimental): Participants met in groups for 2 hours thrice weekly (M/W/F). During the first hour, the counselor facilitated discussion of 1 of the 12 RBT module topics, repeated three times during the course of the 12-week intervention (as in RBT). A patient-led group served the purpose of mutual support during the second hour. The counselor facilitated but did not have direct discussion in these latter groups. The four WHC modules were incorporated into the RBT sessions.
  Interventions: Behavioral: Experimental
- Psycho-education (Active Comparator): Participants met in groups for 2 hours thrice weekly (M/W/F). During the first hour, the counselor facilitated discussion of 1 of the 12 RBT module topics, repeated three times during the course of the 12-week intervention (as in RBT). A patient-led group served the purpose of mutual support during the second hour. The counselor facilitated but did not have direct discussion in these latter groups.
  Interventions: Behavioral: Psycho-education

INTERVENTIONS:
Behavioral: Psycho-education — Receive RBT education and peer-support in a group format.
  Arms: Psycho-education
Behavioral: Experimental — Receive RBT education and a pro-active counseling method
  Arms: RBT+WHIC

SUMMARY:
The purpose of this study was to develop and initially evaluate an efficacious, comprehensive, culturally sensitive, women-centered model of care for pregnant South African women by adapting and refining PI Jones' Reinforcement-Based Treatment (RBT) model, at the same time integrating into it the HIV prevention components of Co-I Wechsberg's Women's Health CoOp (WHC) model, yielding an integrated treatment and prevention model, RBT+WHC.

DETAILED DESCRIPTION:
Cape Town is a striking example of the need for women-specific substance abuse treatment, as it is experiencing a devastating level of methamphetamine use (7% of the adult population),especially among women of childbearing age. The use of methamphetamine (hereafter referred to as "meth") is higher in Cape Town than anywhere else in the country. Consequently, there has been a critical need to develop and test a woman-focused intervention that reduces meth use in a highly vulnerable population of South African women.

Since 2001, the Women's Health CoOp (WHC; PI Wechsberg; RO1s DA011609S; AA014488; HD058320) has successfully adapted an evidence-based intervention to reduce sex- and drug-risk behaviors in drug-using South African women. However, with a rapid rise in meth use, the Western Cape is experiencing a new drug epidemic. A previous WHC study data indicated that the WHC had limited success in reducing the use of this among women. Alarmingly, among WHC participants, a greater proportion of pregnant than non-pregnant women reported using meth (n=24/26=92%; n=238/356=67%; p=.01). These findings are underscored by a lack of a focused and intensive treatment for meth-using pregnant women who live in impoverished townships. Thus, this project responded to PA-09-021 International Research Collaboration on Drug Abuse and Addiction Research (R21) by developing treatment options for meth use among pregnant women and using the long collaboration between WHC staff and local treatment providers to develop our first project to treat meth use in pregnant women.

The goal of this project was to develop and initially evaluate an efficacious, comprehensive, culturally sensitive, women-centred model of care for pregnant South African women by adapting and refining PI Jones' Reinforcement-Based Treatment (RBT) model, at the same time integrating into it the HIV prevention components of Co-I Wechsberg's Women's Health CoOp (WHC) model, yielding an integrated treatment and prevention model, RBT+WHC.

The study had two sequential aims: Aim 1: Adapt and pretest a comprehensive drug abuse treatment model, RBT, which integrated the evidence-based WHC HIV prevention model, to produce a comprehensive, culturally sensitive, woman-focused intervention for meth-using pregnant Coloured women, RBT+WHC. Aim 2: Conduct a small-scale randomized controlled trial (RCT) with pregnant Coloured women to determine the acceptability, feasibility, and initial efficacy of the RBT+WHC model relative to a psycho-educational control condition in terms of their respective impact on maternal outcomes, including (a) meth use, (b) frequency of unprotected sex acts, and (c) number of prenatal care visits; and neonatal outcomes including (d) length of hospital stay, (e) birth weight, and (f) gestational age at delivery. About 300 women were screened for the study but only 32 were found to eligible and completed the study.

The public health impact of this project was far-reaching. RBT+WHC aimed to fill a critical gap in substance use treatment research in a social structure where women are disproportionately disenfranchised from receiving healthcare compared with men. Furthermore, this initial study laid the foundation for a full-scale RCT to examine the impact of RBT+WHC on an array of maternal and neonatal outcomes, within the population of pregnant Coloured as well as Black and White South African women.

ELIGIBILITY:
Inclusion Criteria:

* are 18 years of age or older
* self-identify as "Coloured" (this is a cultural grouping of people with mixed-race ancestry)
* live in the Cape Town township communities of Mitchell's Plain, Delft, Elsie's River, Belhar, Bishop Lavis, or Ravensmead
* meet current DSM-IV criteria for methamphetamine abuse or dependence
* are willing to enter drug abuse treatment
* report unprotected sex in the past 30 days
* are HIV negative
* provide verifiable locator information for follow-up interview
* are 20-28 weeks pregnant, inclusive, and determined by last menstrual period

Exclusion Criteria:

* are male
* are younger than 18 years
* do not self-identify as "Coloured"
* do not live in the Cape Town township communities of Mitchell's Plain, Delft, Elsie's River, Belhar, Bishop Lavis, or Ravensmead
* do not meet current DSM-IV criteria for methamphetamine abuse or dependence
* are not willing to enter drug abuse treatment
* have not reported unprotected sex in the past 30 days
* are HIV positive
* do not provide verifiable locator information for follow-up interview
* are not 20-28 weeks pregnant
* are not able to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Methamphetamine practices | 3 months after randomization
  Frequency of methamphetamine use in past 30 days measured by RRBA (WHC Revised Risk Behavior Assessment) and urine test
Prenatal care | At time of delivery
  Number of prenatal care visits measured by chart review of hospital record
Length of hospital stay | At time of delivery
  Length of hospital stay measured by chart review of hospital record

SECONDARY OUTCOMES:
Drug Use | 3 months after randomization
  Frequency of opioid, cocaine, mandrax, marijuana, and self-report nicotine use in past 30 days measured by RRBA (WHC Revised Risk Behavior Assessment) and urine test
Drug and alcohol use composite scores | 3 months after randomization
  Drug and alcohol composite scores measured by the Addiction Severity Index
Alcohol use | 3 months after randomization
  Frequency of alcohol use in past 30 days measured by RRBA and breath test
Sexual practices | 3 months after randomization
  Frequency of unprotected sexual acts at last sexual encounter and in past 30 days measured by RRBA
Birthweight | At time of delivery
  Birthweight measured by chart review of hospital record
Estimated gestational age | At time of delivery
  Estimated gestational age measured by chart review of hospital record

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Browne, ScD, Principal Investigator — RTI International
Locations (1):
- Medical Research Council, Tygerberg, Western Cape, South Africa